CLINICAL TRIAL: NCT02081755
Title: A 36 Month Multi-center, Open Label, Randomized, Comparator Study to Evaluate the Efficacy and Safety of Everolimus Immunosuppression Treatment in Liver Transplantation for Hepatocellular Carcinoma Exceeding Milan Criteria
Brief Title: Safety and Efficacy of Everolimus Treatment in Liver Transplantation for Liver Cancer
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013-307
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Immunosuppressive Agents; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus; Tacrolimus; Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus and Tacrolimus (Experimental): Everolimus Dosing: 1.5 mg BID (3.0 mg/day) Tacrolimus Dosing: 0.05 mg/kg BID
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Tacrolimus and Myfortic or CellCept or Imuran (Active Comparator): Myfortic: 360 mg to 1080 mg BID OR CellCept: 500 mg to 1500 mg BID OR Imuran: 0.5mk/kg to 2mg/kg QD AND Tacrolimus Dosing: 0.05 mg/kg BID
  Interventions: Drug: Tacrolimus; Drug: Myfortic; Drug: CellCept; Drug: Imuran

INTERVENTIONS:
Drug: Everolimus — Everolimus Dosing: 1.5 mg BID (3.0 mg/day) for 12 months
  Other Names: Zortress; Afinitor
  Arms: Everolimus and Tacrolimus
Drug: Tacrolimus — Tacrolimus Dosing: 0.05 mg/kg BID for 12 months
  Other Names: Prograf
Drug: Myfortic — Myfortic®: 360 mg to 1080 mg BID for 12 months
  Other Names: Mycophenolic Acid
  Arms: Tacrolimus and Myfortic or CellCept or Imuran
Drug: CellCept — CellCept: 500 mg to 1500 mg BID for 12 months
  Other Names: Mycophenolate Mofetil
  Arms: Tacrolimus and Myfortic or CellCept or Imuran
Drug: Imuran — 0.5 mg/kg to 2 mg/kg QD for 12 months
  Other Names: Azathioprine
  Arms: Tacrolimus and Myfortic or CellCept or Imuran

SUMMARY:
This study is a prospective Phase IV study to determine if the use of Everolimus results in lower liver tumor recurrence and improved patient and graft survival after liver transplant for hepatocellular carcinoma (HCC). The immunosuppressive comparators will be Everolimus and Tacrolimus therapy compared to Tacrolimus and Mycophenolic acid/Mycophenolate Mofetil/Azathioprine. Primary outcomes data is disease free survival (the time from randomization to HCC recurrence or death). Secondary outcomes are rate of recurrence of Hepatitis C, problems related to wound healing, hernia repair within the first 12 months, hepatic arterial thrombosis, renal function, acute cellular rejection, post-transplant diabetes, hypertension, and hyperlipidemia.

DETAILED DESCRIPTION:
The study population will consist of approximately 336 patients (224 Everolimus and Tacrolimus and 112 Tacrolimus and Mycophenolic acid/Mycophenolate Mofetil/Azathioprine). Initial screening criteria will include the presence of hepatocellular carcinoma in patients 18 years or older who are candidates to receive a primary orthotopic liver transplant (from deceased or living donor). Within 7 - 12 days post-transplant, patients will be re-evaluated for eligibility for randomization. The criteria include: pre-transplant imaging that shows HCC disease exceeding Milan criteria; pathology review for tumor burden and/or presence of microvascular invasion; AFP >200IU/mL; pre-transplant ablation or resection with HCC recurrence; progression or new tumors; evaluation to rule out any hepatic vessel complication.

Subjects will remain in study treatment until Month 12 at which time the subject and investigator will determine the preferred immunosuppressive regimen. Subjects will be followed for an additional 24 months for outcome data as described above.

ELIGIBILITY:
Screening Inclusion Criteria:

* Have a diagnosis of hepatocellular carcinoma (HCC) and high risk for HCC recurrence
* Able to provide written informed consent
* Male and female patients of any race, 18 years or older
* De novo recipients of a primary orthotopic liver transplant from a deceased or living donor
* Patients willing to comply with study requirements
* Women of child-bearing potential (WOCBP) must agree to use an effective method(s) of contraception during treatment and during the post treatment follow-up period

Screening Exclusion Criteria:

* Past or present malignancy within the last 5 years.
* Severe infection considered by the local site investigator to be unsafe for study participation.
* Use of other investigational drugs at the time of screening or within the last 30 days.
* Patients scheduled for a combined transplant (such as liver-kidney), or having a previous solid organ, bone marrow, or autologous islet cell transplant.
* Recipients of donor/recipient ABO incompatible grafts.
* Recipients of organs from human immunodeficiency virus (HIV) or HBsAg positive donors.
* Macrovascular tumor invasion.
* Proteinuria greater than 2 grams/24 hours.
* Conditions which can result in impaired absorption, distribution, metabolism or excretion of the study treatment.
* Patients with non-infectious pneumonitis.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Women of child-bearing potential (WOCBP) not practicing an effective method(s) of contraception.
* Patients who receive sirolimus (Rapamune®) as part of their transplant immunosuppression regimen

Randomization Screening Inclusion Criteria :

- For patients with a history of any hepatic vessel thrombosis, occlusion, stent placement, or major revision of liver vessels, must have a Doppler ultrasound prior to randomization to rule out any hepatic vessel complication, including hepatic arterial thrombosis (HAT).

Randomization Exclusion Criteria:

* Patients who receive sirolimus (Rapamune) any time prior to randomization will be withdrawn from the study.
* Patients who develop clinically significant systemic infections requiring active use of IV antibiotics any time prior to randomization.
* Wound healing problem, per Investigator's assessment, that would make the patient ineligible for study randomization
* Confirmed presence of a thrombosis in a major hepatic artery(s), major hepatic vein(s), portal vein or inferior vena cava via Doppler ultrasound or other imaging obtained prior to randomization.
* Proteinuria greater than 2 grams/24 hours.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive everolimus or be randomized into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) defined as the time from randomization to the time of tumor recurrence or death, whichever occurs first. | Through Month 36

SECONDARY OUTCOMES:
Tumor recurrence sites | Through Month 36
Hepatitis C recurrence rate | Through Month 36
Renal function | Through Month 36
Acute cellular rejection | Through Month 36
Post-transplant diabetes | Through Month 36
Hypertension | Through Month 36
Hyperlipidemia | Through Month 36
Wound healing and associated risk factors | Through Month 36
Hernia repair | Through Month 36
Hepatic arterial thrombosis | Through Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Goran Klintmalm, MD, PhD, Principal Investigator — Baylor Health Care System
Locations (9):
- United States (9):
  - University of California at San Francisco, San Francisco, California
  - Northwestern University School of Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Tennessee- Methodist University Hospital, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No